CLINICAL TRIAL: NCT05727072
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Investigate Safety, Tolerability, and Pharmacokinetics With Single Intravenous Ascending Doses and Single and Multiple Subcutaneous Doses of LY3848575 in Healthy Participants, Including First-generation Japanese Participants
Brief Title: A Study of LY3848575 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18589; J4F-MC-CYAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3848575 IV (Experimental): Single ascending doses of LY3848575 administered intravenously (IV).
  Interventions: Drug: LY3848575
- Placebo IV (Placebo Comparator): Placebo administered IV.
  Interventions: Drug: Placebo
- LY3848575 SC (Experimental): Multiple doses of LY3848575 administered subcutaneously (SC).
  Interventions: Drug: LY3848575
- Placebo SC (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3848575 — Administered IV.
  Arms: LY3848575 IV
Drug: LY3848575 — Administered SC.
  Arms: LY3848575 SC
Drug: Placebo — Administered IV.
  Arms: Placebo IV
Drug: Placebo — Administered SC.
  Arms: Placebo SC

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3848575 when administered either intravenously or subcutaneously in single ascending or multiple doses in healthy non-Japanese and first generation Japanese participants. The study will also assess how fast LY3848575 gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants. The study will last up to approximately 142 days excluding the screening period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Have body weight of at least 50 kilograms (kg) for males and 40 kg for females, and body mass index of 18 to 30 kilograms per meter squared (kg/m²), inclusive
* For cohorts with Japanese participants: To qualify as a participant of the first-generation Japanese origin, the participant, the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan

Exclusion Criteria:

* Are currently enrolled in any other clinical study involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have participated, within the last 3 months, in a clinical study involving an IP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through 142 days
  A summary of TEAEs, SAEs and Other Non-serious Adverse Events (AEs), Regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3848575 When Administered IV. | End of infusion through day 85
  PK: AUC of LY3848575 When Administered IV.
PK: AUC of LY3848575 When Administered SC. | Predose through day 85
  PK: AUC of LY3848575 When Administered SC.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No